CLINICAL TRIAL: NCT00006435
Title: Natural History of Plexiform in Neurofibromatosis Type I
Brief Title: Study of Plexiform Neurofibromas in Neurofibromatosis Type 1
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010027; 01-C-0027; NCT00445991 (obsolete NCT alias)
Record Dates: First submitted 2000-11-03; First posted 2000-11-06 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Plexiform Neurofibromas; NF1
Keywords: Tissue Repository; Growth Rate; Volumetric MRI
MeSH Terms: conditions — Neurofibroma, Plexiform

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

-Plexiform neurofibromas in patients with NF1 are a significant cause of morbidity but little is known about the natural history of these lesions.

Objectives:

* The purpose of this study is to monitor the natural history of plexiform neurofibromas and to evaluate the usefulness of volumetric MRI tumor measurements in this disease.
* Other goals of the study are to provide a body of normative data on the growth rate of plexiform neurofibromas and to establish a tissue repository and pathology review center to allow future studies of the pathogenesis of neurofibromas and clinical trials of potential therapeutic agents.

Design

- This study is coordinated by Dr. Bruce Korf, and was initiated when he was at the Partners Center for Human Genetics, Boston, MA.

DETAILED DESCRIPTION:
Background:

-Plexiform neurofibromas in patients with NF1 are a significant cause of morbidity but little is known about the natural history of these lesions.

Objectives:

* The purpose of this study is to monitor the natural history of plexiform neurofibromas and to evaluate the usefulness of volumetric MRI tumor measurements in this disease.
* Other goals of the study are to provide a body of normative data on the growth rate of plexiform neurofibromas and to establish a tissue repository and pathology review center to allow future studies of the pathogenesis of neurofibromas and clinical trials of potential therapeutic agents.

Design

- This study is coordinated by Dr. Bruce Korf, and was initiated when he was at the Partners Center for Human Genetics, Boston, MA.

ELIGIBILITY:
* INCLUSION
* Diagnosis of Neurofibromatosis: All study subjects will fulfill two or more of the diagnostic criteria listed below for NF1.

  * Six or more caf(SqrRoot)(Copyright)-au-lait macules

    * 1.5cm or larger in postpubertal individuals
    * 0.5 cm or larger in prepubertal individuals
  * Two or more neurofibromas of any type or 1 or more plexiform neurofibroma
  * Freckling in the axilla or groin
  * Optic glioma (tumor of the optic pathway)
  * Two or more Lisch nodules (benign iris hamartomas)
  * A distinctive bony lesion

    * Dysplasia of the sphenoid bone
    * Dysplasia or thinning of long bone cortex
  * A first degree relative with NF-1
* Plexiform Neurofibroma: A plexiform neurofibroma fulfilling entry criteria for the study will be defined as a diffuse soft tissue or nerve enlargement in a patient with NF1 that is causing, or has potential to cause, disfigurement or functional disability.
* Distribution of Plexiform Neurofibromas by site: A total of 300 plexiform neurofibromas will be studied, consisting of 100 tumors in the following three groups (based on region of maximal involvement):

  * Head and Neck
  * Trunk and Limbs (externally visible)
  * Trunk and Limbs (internal) [spinal plexiform neurofibromas involve two or more levels with connection between the levels or extending laterally along the nerve]
* Subject Ascertainment: Study subjects will be ascertained at any of the participating clinical centers. It is expected that these will include subjects already followed in these clinics, as well as newly diagnosed patients

EXCLUSION

* Presence of metallic implant(s) that will make the patient unable to have MRI studies
* Presence of medical or psychological condition that will make the patient unable to tolerate MRI studies or anesthesia (if needed)
* Inability to image tumor or define tumor margins by MRI (which may be determined after the initial study)
* Failure to obtain initial MRI within 60 days of enrollment
* Previous radiation therapy to site of plexiform neurofibroma
* Surgery involving the plexiform neurofibroma (excluding biopsy) within a six month period before enrollment
* Current antineoplastic therapy
* Entry of more than one member of the same family into the study is not permitted

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 300 plexiform neurofibromas will be studied, consisting of 100 tumors in the head/neck and trunk/limbs (externally visible and internal)
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2001-05-18 (Actual); Primary Completion 2007-09-07 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Monitor natural history of plexiform neurofibromas | 3 years
  Monitor natural history of plexiform neurofibromas
Usefulness of volumetric MRI measurements | 4 years
  Usefulness of volumetric MRI measurements

SECONDARY OUTCOMES:
Establish tissue repository & pathology reviews center | 3 years
Body of data regarding growth rate of plexiform neurofibromas | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-C-0027.html